CLINICAL TRIAL: NCT02177435
Title: An Eight Week Randomized, Double-Blind Study Comparing a Fixed Dose Combination of Telmisartan 80 mg Plus Hydrochlorothiazide 12.5 mg to Telmisartan 80 mg in Patients Who Fail to Respond Adequately to Treatment With Telmisartan 80 mg.
Brief Title: Telmisartan With or Without Hydrochlorothiazide in Patients With Mild-to-moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.261
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; telmisartan, hydrochlorothiazide drug combination

ARMS (2):
- Telmisartan plus Hydrochlorothiazide (Experimental)
  Interventions: Drug: Telmisartan/Hydrochlorothiazide; Drug: Placebo
- Telmisartan (Experimental)
  Interventions: Drug: Telmisartan; Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan
Drug: Telmisartan/Hydrochlorothiazide
  Arms: Telmisartan plus Hydrochlorothiazide
Drug: Placebo

SUMMARY:
Study to demonstrate that a fixed dose combination of telmisartan 80 mg plus hydrochlorothiazide (HCTZ) 12.5 mg (FDC 80/12.5) is superior to telmisartan 80 mg (Telm 80) alone in patients who failed to respond adequately to Telm 80 monotherapy in lowering seated trough diastolic blood pressure (DBP) after eight weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* History of mild-to-moderate hypertension
* Patients who fail to respond adequately to telmisartan monotherapy
* Participants between 18 and 80 years of age
* Ability to provide written informed consent

Exclusion Criteria:

* Patients taking more than three anti-hypertensive medications at the screening visit
* Pre-menopausal women (last menstruation ≤ 1 year prior to start of screening)

  * Who are not surgically sterile (hysterectomy, tubal ligation)
  * Who are NOT practicing acceptable means of birth control or who do NOT plan to continue using an acceptable method throughout the study
* Any women:

  * Who has a positive serum pregnancy test at screening (Visit 1) or baseline (Visit 4)
  * Who is nursing
* Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

  * SGPT (ALT) (serum glutamate pyruvate transaminase) or SGOT (AST) (serum glutamate oxaloacetate transaminase) greater than two times the upper limit of normal
  * Serum creatinine > 2.3 mg/dL
* Clinically relevant sodium depletion, hyperkalemia, or hypokalemia at baseline
* Known or suspected secondary hypertension
* Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney; post-renal transplant patients, presence of only one functioning kidney
* Congestive heart failure (CHF) (NYHA (New York Heart Association) class CHF III-IV)
* Unstable angina within the past three months
* Stroke within the past six months
* Myocardial infarction or cardiac surgery within the past three months
* PTCA (percutaneous transluminal coronary angioplasty) within the past three months
* History of angioedema
* Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator
* Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
* Administration of digoxin or other digitalis-type drugs
* Patients with insulin treated Type II diabetes mellitus whose diabetes has not been stable and controlled for at least the past three months as defined by an HbA1C ≥ 10%
* Known drug or alcohol dependency within the past one year period
* Concomitant administration of medications known to affect blood pressure, except medications allowed by the protocol
* Patients receiving any investigational therapy within one month of signing the informed consent form. Patients who have participated in previous telmisartan studies may participate in this study provided there has been at least one month between discontinuing the previous study and signing the consent for the present study
* Known hypersensitivity to any component of the formulations
* Any clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of trial medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 1999-02; Primary Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in seated diastolic blood pressure (DBP) at trough | Baseline (day 0), day 28, day 56

SECONDARY OUTCOMES:
Change from baseline in seated systolic blood pressure (SBP) at trough | Baseline (day 0), day 28, day 56
Change from baseline in standing DBP and SBP at trough | Baseline (day 0), day 28, day 56
Blood pressure control (seated DBP < 90 mmHg) | 16 weeks
Systolic blood pressure response | 16 weeks
Number of patients with abnormal findings in physical examination | Baseline (screening), day 0 and day 56
Changes from baseline in heart rate | Baseline (screening), day -56, -28, 0, 28 and 56
Number of patients with abnormal changes in laboratory parameters | Baseline (screening), day 0 and day 56
Number of patients with abnormal changes in resting 12-lead ECG (electrocardiogram) | Baseline (screening), day 0 and day 56
Orthostatic changes in blood pressure | Baseline (screening), day -56, -28, 0, 28 and 56
Number of patients with adverse events | up to 16 weeks